CLINICAL TRIAL: NCT06217601
Title: Impact Evaluation of the Digital Connect Project for Homebound Older Adults: A Target Trial Emulation
Brief Title: Impact Evaluation of the Digital Connect Project for Homebound Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Digital Connect
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Aging Well
Keywords: Ageing; Digital intervention; Functional capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment status (Experimental): To account for immortal time bias, each subject will be created with two clones at time zero and assigned each of the two clones to either treatment or no-treatment status, respectively. The treatment status in each evaluative endpoint (i.e., 3-month, 6-month, and 12-month) is defined as subjects who have received the digital intervention for the respective length of time since the time zero during which the intervention has just commenced.
  Interventions: Behavioral: Digital intervention through Tablet
- No-treatment status (Placebo Comparator): To account for immortal time bias, each subject will be created with two clones at time zero and assigned each of the two clones to either treatment or no-treatment status, respectively. The corresponding no-treatment status is defined as subjects who have not received the digital intervention for the corresponding length of time.
  Interventions: Behavioral: Digital intervention through Tablet

INTERVENTIONS:
Behavioral: Digital intervention through Tablet — Web-based multi-domain lifestyle training intervention will be conducted to promoted and focus three lifestyles: nutritional advice, exercise and cognitive training; chat communication with research team, and personalized agenda on daily activities and an information library.

SUMMARY:
The goal of this study is to evaluate the impact of the Digital Connect Project on increasing functional capacity defined by the WHO-ICOPE and health-related quality of life (HRQL) among homebound older adults.

DETAILED DESCRIPTION:
The Hong Kong Jockey Club Charities Trust is launching the Digital Connect project to increase the well-being and social connectedness of the homebound older adults. A total of 32 NGOs are applying for 7,500 tablets and data plan (in total) through this project. Different digital programs will be rolled out to enhance their well-being and social connectedness. This study aim is to capture the impact of this Digital Connect project on the health outcomes of the homebound older adults. The tablet intervention will be offered by the NGOs within a 2-year timeframe. Web-based multi-domain lifestyle training intervention will be conducted to promoted and focus three lifestyles: nutritional advice, exercise and cognitive training; chat communication with research team, and personalized agenda on daily activities and an information library.

The object of this study is to explore the dose-response relationship between online engagement in the different types of activity and the improvement in the corresponding health outcomes, including the five domains: (1) Physical function, (2) Cognitive function, (3) Psychological function, (4) Social function and (5) Health-related quality of life. One baseline assessment and four follow-ups will be arranged in every 3-month interval. To account for immortal time bias, each subject will be created with two clones at time zero and assigned each of the two clones to either treatment or control group, respectively.

The engagement experience will be explored by interviewing the participants and service stakeholders through the planning and delivery of the digital intervention for the homebound older adults.

ELIGIBILITY:
Inclusion Criteria:

* age > 65
* consent to participate
* able to participate in the impact assessment as evidence by a test score of > 6 on the Abbreviated Mental Test
* has the functional ability to engage in the digital intervention

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1024 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQL) | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measure by EQ-5D-5L (range from -0.59 to 1.0), higher score indicates better quality of life
Physical function | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measured by Short Physical Performance Battery (range from 0 to 12), with higher score indicating better physical performance
Cognitive function score | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measured by 5-minute Montreal Cognitive Assessment (MoCA) (range from 0 to 30), A score of 26 or over is considered to be normal.
Subjective Memory Score | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measured by 7-item Memory Complaint Scale (MCS) (range from 0 to 14), lower score indicates better memory performance. No MCs (0-2), Mild MCs (3-6), Moderate MCs (7-10), Severe MCs (11-14).
Loneliness score | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measured by 3-item UCLA Loneliness Scale (range 3-9), higher score indicates greater loneliness.
Depression score | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measured by The 8-item Geriatric Depression Scale (range 0 to 8), with higher score indicating higher risk of depression
Social function | Changes from baseline to 3 month, 6 month, 9 month, and 12 month post-intervention.
  Measured by 8-item Social Connectedness Scale Revised (range 0 to 48), <22 indicates lack of social connectedness

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers.